CLINICAL TRIAL: NCT02663258
Title: An Explorative Phase II Study of Anti-PD-1 (Pembrolizumab) Therapy in Metastatic Melanoma (ADAPTeM)
Brief Title: A Study of Anti-PD-1 (Pembrolizumab) Therapy in Metastatic Melanoma (ADAPTeM)
Acronym: ADAPTeM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4254
Record Dates: First submitted 2016-01-12; First posted 2016-01-26 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2016-01

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab arm (Experimental): All participants treated with Pembrolizumab, 200mg iv, 3weekly
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: Keytruda

SUMMARY:
Abbreviated Title: An explorative Phase II study of Anti-PD-1 (Pembrolizumab) in patients with advanced melanoma (ADAPTeM)

Trial Phase: Phase II

Clinical Indication: Stage III unresectable/stage IV metastatic melanoma

Trial Type: Exploratory Phase II trial

Route of administration: Intravenous Pembrolizumab, 200mg, 3weekly

Trial Blinding: Unblinded; open label Phase II study

Treatment Groups: All participants treated with Pembrolizumab, 200mg iv, 3weekly

Number of trial subjects: 40

Estimated duration of trial: 24 months

Duration of Participation: 24 months

DETAILED DESCRIPTION:
This is a single arm, single agent, open label, exploratory translational research study in patients with unresectable stage III or stage IV melanoma being treated with Pembrolizumab. Suitable patients will undergo serial surgical core biopsies (nonradiological) of subcutaneous or lymph node metastases (as judged by an Oncological Surgical Consultant). As a primary endpoint, the investigators will assess the safety and feasibility of undergoing these biopsies within the patient cohort. A total of forty patients will be recruited over a period of two years.

Patients who have provided consent and satisfied the eligibility criteria will undergo baseline CT scanning and peripheral blood sampling. At baseline, biopsies of suitable metastatic lesions will be undertaken and samples sent for histopathological assessment and analysis of molecular and immune parameters. Participants will be treated with Pembrolizumab, 200mg, intravenously, every 3 weeks. At 6 weeks following commencement of Pembrolizumab therapy, a further biopsy or excision of metastatic disease will be performed, unless considered no longer possible on the basis of a near or complete response to treatment. Blood sampling will be performed prior to each cycle and repeat CT scanning will occur every 9 weeks. Response evaluations will be performed according to RECIST 1.1 criteria. Pembrolizumab will be continued as long as study participants are deriving benefit and further biopsies of progressing lesions will be performed where possible.

The investigators aim to evaluate the safety and feasibility of obtaining serial tumour biopsies or excisions of metastatic disease during treatment with Pembrolizumab with exploration of the i) mechanistic activity of Pembrolizumab, ii) identification of intratumoural and peripheral factors limiting response, iii) identification of candidate predictive biomarker panels based on (i) and (ii) and iii) use of circulating free DNA (cfDNA) as a surrogate marker of response and guide to duration of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic melanoma (cutaneous or mucosal)
2. Male or female, 18 years or older
3. Presence of subcutaneous or lymph nodes metastases amenable to surgical core biopsy (as judged by an Oncological Surgical Consultant)
4. Have measurable disease based on Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
5. Have provided tissue from an archival tissue sample or newly obtained core biopsy of a tumour lesion.
6. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
7. Any number of previous lines of treatment for metastatic melanoma including treatment naïve patients.
8. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
11. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Has a known additional malignancy that is progressing or requires active treatment.

   Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule.

   Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CD137 antibody.
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
The percentage of patients that undergo serial core biopsies of metastatic lesions during treatment with Pembrolizumab | At study progression (average of 9 months) or 24 months after last patient enrolled
  The primary endpoint of the study is to assess the feasibility of obtaining sequential tumour biopsies will be achieved when sequential biopsies (at baseline, week 6 and at disease progression), have successfully been carried out in a minimum of 75% of patients (i.e. 29 out of 40).The percentage of patients with complete tumour response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) will be tabulated. Associated 95% CI will be provided for response rates. The duration of objective response (for patients with CR and PR) will be defined as the time from initial CR or PR to the time of disease progression or death (whichever occurs first). For patients who do not die or experience PD, duration of objective response will be censored on the day of the last tumour assessment.

SECONDARY OUTCOMES:
The complication rate associated with undergoing serial core biopsies | At study progression (average of 9 months) or 24 months after last patient enrolled
  Complication rate will be defined as the proportion of patients who have hospital admission due to complication of biopsy e.g. infection/bleeding/pain control and/or delay in Pembrolizumab treatment due to complication of biopsy. This will be presented as a proportion with the 95% confidence interval.
Objective response rate | At study progression (average of 9 months) or 24 months after last patient enrolled
  Objective response rate defined as proportion of patients with a best response of complete response (CR) or partial response (PR).
Progression free survival | At study progression (average of 9 months) or 24 months after last patient enrolled
  Progression-free survival (PFS) will be defined as the time from the first day of Pembrolizumab treatment (cycle 1 day 1) until documented disease progression or death (whichever occurs first). Patients who do not have documented PD or death will be censored on the day of last tumour assessment (last follow-up).
Overall survival | At study progression (average of 9 months) or 24 months after last patient enrolled
  Overall survival will be measured from the first day of treatment until death or last follow-up. Overall survival will be presented graphically using the Kaplan-Meier method. Median time to event and 95% CI will be estimated from the Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: James Larkin, Principal Investigator — Royal Marsden NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No